CLINICAL TRIAL: NCT02292225
Title: A Phase 1b Study of Duvelisib Administered in Combination With Obinutuzumab in Patients With CLL/SLL Previously Treated With a Bruton's Tyrosine Kinase Inhibitor (BTKi) (SYNCHRONY)
Brief Title: Duvelisib With Obinutuzumab in Patients With CLL/SLL Previously Treated With a BTKi (SYNCHRONY)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The scope of the program has been reduced to focus resources on studies which can potentially enable the registration of duvelisib.
Sponsor: SecuraBio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPI-145-18
Record Dates: First submitted 2014-11-10; First posted 2014-11-17 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Lymphocytic Leukemia, Chronic; Lymphoma, Small Lymphocytic
Keywords: Phase 1b, CLL/SLL, PI3K
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Hereditary Sensory and Autonomic Neuropathies | interventions — duvelisib; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IPI-145 in Combination with Obinutuzumab (Experimental)
  Interventions: Drug: IPI-145 (duvelisib); Drug: Obinutuzumab

INTERVENTIONS:
Drug: IPI-145 (duvelisib) — 25mg and/or 5mg oral capsule
  Other Names: Duvelisib
Drug: Obinutuzumab — 1000mg/40mL single-use vials
  Other Names: GAZYVA

SUMMARY:
To evaluate the safety, pharmacokinetics, and pharmacodynamics of Duvelisib (IPI-145) in combination with obinutuzumab in patients with Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma previously treated with a BTKi.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, dose escalation, safety and tolerability study of Duvelisib (IPI-145) in combination with obinutuzumab in subjects with Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma previously treated with a BTKi therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Diagnosis of Chronic lymphocytic leukemia or Small lymphocytic lymphoma that meets at least one of the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria for treatment (Binet Stage ≥ B and/or Rai Stage ≥ I with symptoms)
* Measurable disease with a lymph node or tumor mass >1.5 cm in at least one dimension as assessed by computed tomography (CT)
* Previous exposure to BTKi therapy and meets at least one of the below criteria:

  * Progressive disease while receiving a BTKi therapy, or stable disease as best response after 12 months of receiving a BTKi therapy
  * Discontinued a BTKi therapy due to BTKi treatment-related intolerance
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (corresponds to Karnofsky Performance Status [KPS] ≥60%)
* Subjects must be able to receive outpatient treatment and laboratory monitoring (where specifically indicated) at the institution that administers study drug for the entire treatment period

Exclusion Criteria:

* Richter's transformation or prolymphocytic leukemia
* Refractory to obinutuzumab (defined as progression or relapse <12 months of receiving obinutuzumab monotherapy or <24 months of receiving an obinutuzumab-containing regimen)
* Progressive disease while previously receiving a PI3K inhibitor (e.g. GS-1101 [idelalisib], duvelisib) or a serious/severe AE related to PI3K inhibitor treatment
* History of severe reaction to prior monoclonal antibody therapy (defined as a Grade 4 event and/or requiring permanent discontinuation)
* Human immunodeficiency virus (HIV) or Human T Cell Lymphotropic Virus 1 (HTLV-1) infection
* Prior, current, or chronic hepatitis B or hepatitis C infection
* History of tuberculosis treatment within the preceding 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-02; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) | 28 days
Treatment-emergent adverse events (TEAEs) | Up to 30 days from last dose of study treatment

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to 2 years from the first dose of study treatment
Duration of response (DOR) | Up to 2 years from the first dose of study treatment
Progression-free survival (PFS) | Up to 2 years from the first dose of study treatment
Overall survival (OS) | Up to 2 years from the first dose of study treatment or until study treatment is completed, whichever is later
BTK mutation status | Baseline
Pharmacokinetic (PK) parameters of duvelisib and IPI-656 (major metabolite) | Week 1, Week 2, Months 2, 4, 7, 11, 15, 19

CONTACTS AND LOCATIONS:
Locations (7):
- United States (6):
  - La Jolla, California
  - Boston, Massachusetts
  - Hackensack, New Jersey
  - New Hyde Park, New York
  - Columbus, Ohio
  - Houston, Texas
- Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No